CLINICAL TRIAL: NCT00263237
Title: A Pilot Study of Safety and Efficacy of the Oral IL-12/23 Inhibitor, STA-5326 Mesylate, for Symptomatic Gastrointestinal Inflammation Associated With Common Variable Immunodeficiency
Brief Title: STA-5326 Meslylate to Treat Gut Inflammation Associated With Common Variable Immunodeficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060037; 06-I-0037
Record Dates: First submitted 2005-12-07; First posted 2005-12-07 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-07-23

CONDITIONS: Common Variable Immunodeficiency
Keywords: T Cell; Lymphocyte; Lamina Propria; Malabsorption; Colonoscopy; Common Variable Immunodeficiency; CVID; Gastrointestinal Inflammation
MeSH Terms: conditions — Common Variable Immunodeficiency; Malabsorption Syndromes | interventions — apilimod

INTERVENTIONS:
Drug: STA-5326

SUMMARY:
This study will determine whether an experimental medicine, STA-5326 mesylate, is safe to use in patients with common variable immunodeficiency (CVID) who have inflammation of the gut. It will also determine if patients who take this drug show improvement in their symptoms, decrease in inflammatory chemicals in the gut, changes in their immune cells, and improvement in how their gut is functioning to absorb food.

Patients between 18 and 75 years of age with CVID and chronic diarrhea or involuntary weight loss of more than 5 percent of their past body weight over the past 12 months may be eligible for this study. Candidates are screened with a review of their medical records, a medical history and physical examination, blood, urine and stool tests, chest x-rays and skin test for exposure to tuberculosis, and a hydrogen breath test. For the latter, breath samples are collected before and every 20 minutes (for 2 hours) after the subject drinks a sugar solution. This test determines the digestive effects of bacteria in the upper intestine. Samples are collected by having the subject blow into a balloon.

Participants undergo the following tests and procedures:

Immune System and Gastrointestinal Evaluation

* 48-hour stool fat collection (measures the amount of undigested fat in the stool): Subjects keep a diary of what they eat for a 48-hour period. At the beginning of the 48 hours they take two dye capsules and then take another two capsules 48 hours later. They collect a stool sample when they pass the second set of capsules in their bowel movement. An additional 24-hour stool collection is tested for loss of protein in the stool.
* D-xylose absorption test (measures the ability of the gut to absorb nutrients): Subjects drink a solution of d-xylose (a sugar substitute). Blood samples are collected before and 1 hour after drinking the solution.
* Upper endoscopy: A thin flexible lighted tube is advanced through the mouth to evaluate the esophagus, stomach and beginning of the small intestine.
* Lower endoscopy: A thin flexible lighted tube is advanced through the rectum to evaluate the colon.

Treatment Period (Study days 1 to 57)

* Physical examination - study days 1, 8, 15, 29, 43 and 57
* Blood samples to test the levels of STA-5326 in the blood. On study days 1 and 57, samples are collected before the medication dose and 1, 2, 4, 6 and 8 hours after the dose; on day 29, one sample is collected before the medication dose.
* Blood samples for routine safety testing - study days 1, 8, 15, 29, 43 and 57
* Medication history - study days 1, 8, 15, 29, 43 and 57
* Interview about pain, discomfort, and well being - study days 1, 8, 15, 29, 43 and 57
* Pregnancy test for women who can become pregnant - study days 15, 43, and 57
* D-xylose absorption test - study days 29 and 57
* Electrocardiogram - study days 29 and 57
* Urine test - study days 29 and 57
* Blood test for research on immune cells - study day 57
* Repeat endoscopies and studies of gut function (24- and 48-hour stool collections)

Follow-up period (Day 85 and day 113)

-Physical examination, blood tests, medication history, questions about pain, discomfort and well being

DETAILED DESCRIPTION:
The purpose of this study is to assess the toxicity of the oral IL-12/23 inhibitor STA-5326 mesylate in subjects with common variable immunodeficiency (CVID) and associated symptomatic gastrointestinal inflammation. Common variable immunodeficiency is a clinically heterogeneous disorder characterized by decreased serum immunoglobulin IgG and IgA levels. In addition to chronic or recurrent pyogenic sino-pulmonary infections, many patients develop non-infectious gastrointestinal manifestations that can be disabling or fatal. Currently there is no standard therapy for the associated gastrointestinal disease outside of empiric nutritional intervention for weight loss and non-specific anti-diarrheal agents.

Recently gut inflammation complicating CVID has been characterized as a Th1 inflammatory response, with excess cytokine production associated with diarrhea and weight loss as well as reduced D-xylose absorption and steatorrhea. This protocol represents the first attempt to test specific anti-IL-12 therapy in this patient group; it has been previously shown that therapy targeted to IL-12/23 successfully treated the Th1 gut inflammation of Crohn's disease. While this protocol is designed to measure the safety of STA-5326 mesylate in CVID patients, it will also measure effects on symptoms, gut function, expression of immune cell surface markers and production of cytokines from blood and gut mucosal mononuclear cells.

CVID patients with gastrointestinal symptoms of malabsorption, maldigestion, and chronic diarrhea will be enrolled into this study. Subjects (up to a total of 10 individuals) will receive STA-5326 mesylate 100 mg per os (PO) once daily (QD) (equivalent to 70 mg STA-5326 free base) for 8 weeks. Subjects will have pretreatment and end-of-study procedures, including upper and lower endoscopies, to measure changes in immune responses and physiologic measures of gut function, as well as routine safety monitoring throughout the treatment period. Variables will include safety (adverse event rate), clinical (weight, stool frequency, results of gut absorption tests), and laboratory (lymphocyte and cytokine assays) parameters for descriptive summary statistical analysis (n, mean, median, standard deviation, minimum and maximum range).

ELIGIBILITY:
* INCLUSION CRITERIA:

A subject is eligible for the study if all of the following criteria are met:

Has given written informed consent prior to screening.

Is male or female aged 18 through 75 years.

Has CVID diagnosed definitively prior to screening (based on the IUIS criteria).

Has a documented, unintended loss of greater than 5% of their body weight over the last year or requires nutritional supplements to maintain his/her body weight OR has chronic diarrhea defined as a complaint of liquid stools for at least 4 consecutive weeks (and an output of greater than 200 g stool/24hr on a diet of at least 1600 calories with 60 g fat.)

If taking oral antibiotics chronically, must have used a stable dose of the antibiotic continuously for at least 2 weeks prior to start of screening period.

Not taking any potential CYP3A4 inhibitors/inducers (e.g., macrolide antibiotics, HIV protease inhibitors, antifungals, grapefruit juice, St. John's Wort).

EXCLUSION CRITERIA:

A subject is excluded from the study if any of the following criteria are met:

General Criteria:

Has any clinically significant disease (e.g., renal, hepatic, neurological, cardiovascular, pulmonary, endocrinologic, psychiatric, hematologic, urologic, or other acute or chronic illness) that in the opinion of the investigator would make the subject an unsuitable candidate for this trial.

Is a woman who has a positive serum pregnancy test or who is breast-feeding.

Is a woman of childbearing potential or a man who does not agree to use two forms of contraception during the course of the study and follow-up period.

Has hypersensitivity to any of the components of STA 5326 mesylate drug product.

Has any of the following clinical chemistry values:

AST greater than 2.5 x upper limit of normal (ULN).

ALT greater than 2.5 x ULN.

Serum bilirubin greater than 1.5 x ULN.

Serum creatinine greater than 1.5 x ULN.

Alkaline phosphatase greater than 2.5 x ULN.

Has a hemoglobin level less than 9 g/dL or hematocrit less than 30%.

Has a Prothromin Time INR greater than 1.3 or a Partial Thromboplastin Time greater than 3 sec compared to control value.

Has the following cell counts (cells/microliter):

Platelet count less than 90,000 or greater than 800,000.

White blood cell count less than 1,500.

Neutrophil count less than 900.

Has a current infection requiring intravenous antibiotics, a serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., pneumonia, septicemia).

Has a history of cancer within the past 5 years, with the exception of excised basal cell carcinoma, squamous cell carcinoma of the skin, or cervical carcinoma in situ.

Had a dependency for any illicit drug, chemical, or alcohol within the past 5 years.

Has a history of active tuberculosis (or a CXR with findings suggestive of old TB infection including calcified nodular lesions, apical fibrosis, or pleural scarring), acute or chronic hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).

Gastrointestinal Criteria:

Has a stool sample positive for gastrointestinal infection during screening.

Has a positive hydrogen breath test

Prior Medication Criteria:

Received parenteral corticosteroids within 1 month prior to receiving study drug. The use of short-term or single-dose corticosteroids as a pretreatment regimen for IVIG is acceptable.

Received any investigational drug within 3 months prior to receiving study drug.

Received cyclosporine, tacrolimus, sirolimus, or mycophenolate mofetil within 2 months prior to receiving study drug.

Received any biological product (e.g., infliximab, adalimumab, natalizumab, etc.) within 3 months prior to receiving study drug.

Ever received treatment with STA-5326 mesylate, anti-IL 12 antibodies, or other specific IL 12 inhibitors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2005-12-02; Study Completion 2008-07-23

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hayes MP, Wang J, Norcross MA. Regulation of interleukin-12 expression in human monocytes: selective priming by interferon-gamma of lipopolysaccharide-inducible p35 and p40 genes. Blood. 1995 Jul 15;86(2):646-50. PMID 7605994
- [Background] DeKruyff RH, Fang Y, Umetsu DT. Corticosteroids enhance the capacity of macrophages to induce Th2 cytokine synthesis in CD4+ lymphocytes by inhibiting IL-12 production. J Immunol. 1998 Mar 1;160(5):2231-7. PMID 9498762
- [Background] Larsson S, Linden M. Effects of a corticosteroid, budesonide, on production of bioactive IL-12 by human monocytes. Cytokine. 1998 Oct;10(10):786-9. doi: 10.1006/cyto.1998.0362. PMID 9811532